CLINICAL TRIAL: NCT07391020
Title: Safety Behavior Fading Intervention for Pathological Worry
Brief Title: Text Message Safety Behavior Fading for Pathological Worry
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005991
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Generalized Anxiety Disorder (GAD); Worrying; Anxiety
Keywords: safety behaviors; worry
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Behavior Fading (Experimental): Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their endorsed worry behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a worry behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day. Participants will also be able to track their progress using daily progress charts that show how their daily total safety behavior use changes throughout treatment.
  Interventions: Behavioral: Safety Behavior Fading for Pathological Worry
- Progressive Muscle Relaxation (PMR) (Active Comparator): Individuals randomly assigned to the PMR condition will receive a total of 4 videos over the course of a month (1 video per week, 15 minutes each) wherein participants will be invited to systematically tense and release different muscle groups in the body in order to build awareness of tension and relaxation.
  Interventions: Behavioral: Progressive Muscle Relaxation (PMR)

INTERVENTIONS:
Behavioral: Safety Behavior Fading for Pathological Worry — Participants are asked to reduce or eliminate safety behaviors via text message reminders, daily checklist, and daily progress chart to monitor progress.
  Arms: Safety Behavior Fading
Behavioral: Progressive Muscle Relaxation (PMR) — Participants are asked watch weekly videos lasting 15 minutes each that walk them through a progressive muscle relaxation exercise.
  Arms: Progressive Muscle Relaxation (PMR)

SUMMARY:
The current study aims to explore the efficacy of a text message-based Safety Behavior Fading Intervention compared to a PMR control condition.

DETAILED DESCRIPTION:
Safety behavior fading intervention procedures will follow methodology previously used in the Cougle Lab. The safety behavior fading intervention is designed to target a decrease or elimination of worry-related safety behaviors.

Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their endorsed worry behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a worry behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day. Participants will also be able to track their progress using daily progress charts that show how their daily total safety behavior use changes throughout treatment. Text messaging will be managed by EZTexting - a service that manages mass texting protocols. The daily reminder will include the following language: "Hi! This is a friendly reminder to avoid using your checklist behaviors. Please tap the link below to access today's checklist: [link to checklist]." Individuals randomly assigned to the PMR condition will receive a total of 4 videos over the course of a month (1 video per week, 15 minutes each) wherein participants will be invited to systematically tense and release different muscle groups in the body in order to build awareness of tension and relaxation.

ELIGIBILITY:
Inclusion Criteria:

- Elevated worry as defined by a score of 60 or higher on the PSWQ.

Exclusion Criteria:

* Score of 59 or lower on the PSWQ
* If applicable, unstable psychiatric medication usage any time over the past 4 weeks
* Failing attention checks in baseline data collection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ; Meyer et al., 1990) | Day 0, Day 28, Day 56
  Self-report scale that measures levels of worry. Scores range from 16 to 80 with higher scores indicating higher levels of worry.
Worry Behaviors Inventory (Mahoney et al., 2016) | Day 0, Day 28, Day 56
  Self-report scale that measures frequency of worry-related safety behavior use. Scores range from 0 to 44 with higher scores indicating more frequent worry-related safety behavior use.
Generalized Anxiety Disorder Scale-7 (GAD-7; Spitzer et al., 2006) | Day 0, Day 28, Day 56
  Self-report scale that measures generalized anxiety symptom severity. Scores range from 0 to 21, with higher scores indicating higher levels of generalized anxiety.
Credibility and Expectancy Questionnaire (Devilly & Borkovec, 2000). | Day 0
  Self-report scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies. Three items are rated on a 1-9 scale and one item is rated on a 0-100 scale with higher scores meaning greater expectancy and credibility.
Theoretical Framework of Acceptability Questionnaire (TFA; Sekhon et al., 2022) | Day 28
  Self-report scale for measuring treatment acceptability. Each item is rated on a 1-5 scale measuring agreement with each statement. For four items, higher scores reflect higher levels of acceptability. For the remaining four items, higher scores reflect lower levels of acceptability. Scores for each subscale range from 4-20.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale-10 (CESD; Andreson, 1994) | Day 0, Day 28, Day 56
  Self-report measure of depression symptom severity. Each item is rated on a 0 to 3 scale. Total scores range from 0 to 30 with higher scores indicating greater depression severity.
NIH Toolbox Fear - Somatic Arousal Scale (Pilkonis et al., 2013) | Day 0, Day 28, Day 56
  Self-report scale measuring levels of anxious somatic arousal. Scores range from 6 to 30, with higher scores indicating higher levels of anxious arousal.
Intolerance of Uncertainty Scale - 12 item version (IUS-12; Carleton et al., 2007) | Day 0, Day 28, Day 56
  Self-report scale that measures intolerance of uncertainty. Scores range from 12 to 60 with higher scores indicating higher levels of intolerance of uncertainty.
Short Scale Anxiety-Sensitivity Index (SSASI; Zvolensky et al., 2018) | Day 0, Day 28, Day 56
  Self-report scale that measures anxiety sensitivity. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Cougle, Ph.D., Study Director — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No